CLINICAL TRIAL: NCT03744494
Title: Comparison of the Therapeutic Efficacy and Patient Satisfaction of Three Techniques of Bilateral Orchidectomy in Prostate Cancer Patients of a Nigerian Sub-population (TEPSO)
Brief Title: Cosmetic Appeal, HRQoL and Effectiveness of Simple and Pseudotesticular Techniques of Orchidectomy in Prostate Cancer
Acronym: TEPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, I.N. Chibuzo, Principal Investigator, University College Hospital, Ibadan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15/0424
Record Dates: First submitted 2018-07-30; First posted 2018-11-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Quality of Life; Orchiectomy
Keywords: orchidectomy; pseudotesticle
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Three groups of patients subjected to a type of orchidectomy each
Who Masked: Participant
Masking Description: The patient, unaware of which surgery was done, would grade the scrotal appearance three months afterwards
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bilateral simple orchidectomy (BSO) (Experimental): The patients would have the testis, epididymis and distal cord structures excised
  Interventions: Procedure: Bilateral simple orchidectomy (BSO)
- Subcapsular orchidectomy (BSCO) (Experimental): The tunica albuginea was incised longitudinally and the testicular parenchyma scraped off it. The hilar region was secured with a haemostat and the parenchyma excised off it. A haemostatic suture was applied at the hilum. A running interlocking water-tight capsular suture was inserted
  Interventions: Procedure: Bilateral Subcapsular Orchidectomy
- Epididymal-sparing orchidectomy (BESO) (Experimental): The epididymal sinus was developed. The epididymal vessels were sequentially clamped and divided, removing the testicle from the epididymis. The caput was looped to meet the head and the adjoining surfaces of the body sutured together (epididymoplasty) Vasectomy done to reduce future risk of epididymitis
  Interventions: Procedure: Bilateral Epididymal-sparing Orchidectomy

INTERVENTIONS:
Procedure: Bilateral simple orchidectomy (BSO)
  Arms: Bilateral simple orchidectomy (BSO)
Procedure: Bilateral Subcapsular Orchidectomy
  Arms: Subcapsular orchidectomy (BSCO)
Procedure: Bilateral Epididymal-sparing Orchidectomy
  Arms: Epididymal-sparing orchidectomy (BESO)

SUMMARY:
The therapeutic efficacy of three types of orchidectomy was ascertained as well as the QoL and scrotal cosmetic satisfaction of patients in the three surgical arms. Two of these surgeries produced a pseudotesticle (BSCO, BESO) while one (BSO) did not.

DETAILED DESCRIPTION:
Patients with prostate cancer (PCa) were grouped into three surgical arms: BSO (bilateral simple orchidectomy), BSCO (bilateral subcapsular orchidectomy) and BESO (bilateral epididymal-sparing orchidectomy). Preoperatively, baseline serum testosterone, PSA, Quality of life (QoL) and pre-operative testicular volumes were obtained. Timed interval sampling for serum testosterone and PSA variation was done post-operatively. By three months post-op, the cosmetic appeal of the scrotal appearance, post-operative pseudotesticular volumes and QoL were also assessed.

The therapeutic efficacy of the surgeries was determined by the rates of decline of serum testosterone and PSA, as well as the nadirs achieved. The variations in the pre-and post-operative QoL was analysed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive consenting patients with histologically confirmed locally advanced or metastatic PCa who have accepted to have an orchidectomy

Exclusion Criteria:

* Patients who have had bilateral orchidectomy
* Those who opt for medical castration

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with advanced prostate cancer
Enrollment: 63 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Summative and domain quality of life scores | Three months
  Expanded Prostate Cancer Index Composite- 26 questionnaires were also used to assess various aspects of the QoL pre-and post-operatively.
  EPIC 26 scores are ranked from 0 to 100 with higher scores indicating better function and less bother. Urinary incontinence, Lower Urinary Tract Symptoms, Bowel function/bother, Sexual function/bother, Hormone and vitality were assessed.
Summative and domain quality of life scores | Three months
  Life Satisfaction -8 questionnaire was used to complement the EPIC-26 in the QoLassessment pre-and post-operatively.
  Lisat-8 is ranked from 1 to 6, with 5 and 6 denoting satisfaction (5: Satisfying; 6: Satisfying) while scores of 4 and below connote varied degrees of dissatisfaction (1: very dissatisfying; 2: Dissatisfying; 3: Rather dissatisfying; 4: Rather satisfying)
  EPIC 26 scores are ranked from 0 to 100 with higher scores indicating better function and less bother. Urinary incontinence, Lower Urinary Tract Symptoms, Bowel function/bother, Sexual function/bother, Hormone and vitality were assessed.
Change in pseudotesticular volume | Three months
  A Prader orchidometer was used to measure the pre-operative testicular volume and post-operative pseudotesticular volume in cm3
Satisfaction with scrotal appearance | three months after the orchidectomy
  Patient rating of cosmetic appeal of the scrotum using a graduated Visual Analog Scale rated between 0 and 100 to signify a score of 0 to 100%. Higher values indicated better satisfaction with scrotal appearance

SECONDARY OUTCOMES:
Serum PSA levels | Three months (timed interval sampling)
  The serum PSA levels in ng/ml were measured pre-operatively, at removal of the testes, hourly for the first three hours, at seven days and three months post-operatively. Percentage PSA declines, PSA nadirs (ng/ml) and time to the attainment of PSA nadirs (hours) were determined from the data obtained.
Serum testosterone levels | Three months (timed interval sampling)
  The serum testosterone levels in nmol/l were measured pre-operatively, at removal of the testes, hourly for the first three hours, at seven days and three months post-operatively. The attainment of surgical castrate levels of 20nmol/l or medical castrate levels of 20 nmol/l or medical castrate levels of 50nmol/l was assessed for as well as the testosterone nadirs achieved (nmol/l) and time to the attainment of testosterone nadirs (hours).

OTHER OUTCOMES:
Socioeconomic standing of the patients | Snap-shot assessment at enrolment
  The EPIC 2.2002 questionnaire was used to determine the relationship, occupational, educational and financial statuses of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Ijeoma NC Chibuzo, MBBS, MSc, Principal Investigator — University College Hospital, Ibadan
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chibuzo INC, Takure AO, Shittu OB, Okeke LI,
- [Derived] Chibuzo INC, Takure AO, Shittu OB, Okeke LI. Cosmetic Appeal, HRQoL, and Effectiveness of Simple and Pseudotesticular Techniques of Orchidectomy in Prostate Cancer. Prostate Cancer. 2021 Nov 26;2021:9968570. doi: 10.1155/2021/9968570. eCollection 2021. PMID 34868687

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03744494/Prot_SAP_ICF_000.pdf